CLINICAL TRIAL: NCT00751959
Title: Surfactant Application During Spontaneous Breathing With CPAP or During Mechanical Ventilation in the Therapy of IRDS in Premature Infants < 27 Weeks
Brief Title: Surfactant Application During Spontaneous Breathing With Continuous Positive Airway Pressure (CPAP) in Premature Infants < 27 Weeks
Acronym: NINSAPP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cologne (Other)
Collaborators: University Hospital Schleswig-Holstein - Lübeck Campus (Unknown); Altona Children's Hospital (Other); Ruhr University of Bochum (Other); Vestische Kinder- und Jugendklinik Datteln (Unknown); Hospital of Leverkusen (Unknown); Kliniken der Stadt Koeln, Kinderkrankenhaus Riehl (Unknown); Heinrich-Heine University, Duesseldorf (Other); Klinikum Aschaffenburg-Alzenau (Other); Asklepios Kliniken Hamburg GmbH (Other); Klinikum Stuttgart (Other); DRK Kinderklinik Siegen (Unknown); University Hospital, Bonn (Other); Charite University, Berlin, Germany (Other); The Clinical Trials Centre Cologne (Other); German Federal Ministry of Education and Research (Other Government)
Responsible Party: Principal Investigator, Angela Kribs, MD, University of Cologne
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Uni-Koeln-439; ISRCTN64011614 (Registry Identifier: ISRCTN)
Record Dates: First submitted 2008-09-11; First posted 2008-09-12 (Estimated); Last update posted 2012-07-19 (Estimated); Status verified 2012-07

CONDITIONS: Respiratory Distress Syndrome, Newborn
Keywords: Continuous positive airway pressure (CPAP); extremely preterm infant; Idiopathic respiratory distress syndrome (IRDS); Surfactant
MeSH Terms: conditions — Respiratory Distress Syndrome, Newborn; Pulmonary Atelectasis | interventions — poractant alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2 (Active Comparator): Conventional therapy with intubation, initiation of mechanical ventilation and surfactant application
  Interventions: Drug: Curosurf
- 1 (Experimental): Surfactant application via a thin endotracheal catheter during spontaneous breathing with CPAP, followed by respiratory support with CPAP
  Interventions: Drug: Curosurf

INTERVENTIONS:
Drug: Curosurf — Surfactant application via a thin endotracheal catheter during spontaneous breathing with CPAP, followed by respiratory support with CPAP
  Arms: 1
Drug: Curosurf — Conventional therapy with intubation, initiation of mechanical ventilation and surfactant application
  Arms: 2

SUMMARY:
This study investigates the efficacy of surfactant application during spontaneous breathing with CPAP in avoiding death and chronic lung disease (CLD) in very immature infants with a gestational age of less than 27 weeks.

DETAILED DESCRIPTION:
80 % of extremely preterm infants with a gestational age of less than 27 completed weeks suffer from severe idiopathic respiratory distress syndrome (IRDS). They are still at high risk of mortality and long term morbidity especially of the lung and the brain. At least death and chronic lung disease (CLD) are related to the need and the duration of mechanical ventilation. Continuous positive airway pressure (CPAP) has been shown to be effective to avoid mechanical ventilation in the treatment of IRDS but it often fails in the most immature infants. Early or prophylactic surfactant application is effective in the treatment of IRDS and is the only causal therapy, but it is usually related to intubation and mechanical ventilation that should be avoided.Therefore to overcome the dilemma between need for mechanical ventilation with surfactant administration on the one hand and surfactant withholding with the use of CPAP on the other hand, a strategy was developed to administer surfactant during spontaneous breathing with CPAP (1). In the proposed prospective randomised controlled trial this strategy shall be compared with the recent gold standard in the therapy of extremely preterm infants with IRDS, that is intubation, mechanical ventilation and surfactant administration. Based on the results of a feasibility (1) study and some clinical observations it is hypothesised that the new approach is superior in avoidance of death and chronic lung disease compared to the recent gold standard.

ELIGIBILITY:
Inclusion Criteria:

* IRDS with Silverman-Score ≥ 5 and / or FiO2 ≥ 0,3
* Postnatal age of more than 10 min. and less than 2 hours
* Gestational age ≥ 23+0 and < 27+0

Exclusion Criteria:

* Primary cardio- pulmonary resuscitation
* Prenatally diagnosed severe malformation
* No parental consent
* Participation in another interventional trial

Ages: 23 Weeks to 26 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 213 (Actual)
Dates: Start 2009-04; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Survival until term without CLD | 13-17 weeks after birth

SECONDARY OUTCOMES:
Survival until term without CLD, IVH>II°, cystic PVL, ROP with need for surgery | 13-17 weeks after birth

CONTACTS AND LOCATIONS:
Overall Officials: Angela Kribs, MD, Principal Investigator — University of Cologne, Clinic for Paediatrics
Locations (13):
- Germany (13):
  - Klinikum Aschaffenburg, Klinik für Kinder- und Jugendmedizin, Aschaffenburg
  - Charité, Berlin
  - Ruhr University of Bochum, Children's Hospital St. Josef Spital, Bochum
  - University Hospital, Dept. of Neonatology, Bonn
  - Kliniken der Stadt Koeln, Kinderkrankenhaus Riehl, Cologne
  - University of Cologne, Clinic for Paediatrics, Cologne
  - Vestische Kinder- und Jugendklinik, Datteln
  - University Hospital, Clinic for Paediatrics, Düsseldorf
  - Asklepios Klinik Barmbek, Hamburg
  - Hospital of Leverkusen, Dept. of Children's Medicine, Leverkusen
  - University Hospital of Schleswig-Holstein, Campus Lübeck, Dept. of Children's Medicine, Lübeck
  - DRK Kinderklinik, Siegen
  - Klinikum Stuttgart, Olgahospital, Stuttgart